CLINICAL TRIAL: NCT06936748
Title: A Study of Spatially Fractionated Radiation Therapy Followed by Sequential Hypofractionated or Conventional Fractionated RT Combined With Iparomlimab and Tuvonralimab for Relapsed and Refractory Bulky Solid Tumors
Brief Title: SFRT+Sequential Hypofractionated/Conventional Fractionated RT+Iparomlimab and Tuvonralimab for Relapsed/Refractory Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-I-2025-014
Record Dates: First submitted 2025-03-26; First posted 2025-04-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Bulky Solid Tumors; Spatially Fractionated Radiation Therapy; Immunotherapy; Iparomlimab and Tuvonralimab
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Combined with Immunotherapy (Experimental): This is a single-arm study. Treatment Protocol Radiotherapy Phase: SFRT: 10-20 Gy/1 fraction to the tumor. Sequential Radiotherapy:Hypofractionated Radiotherapy: 20-70 Gy total (3-12.5 Gy/fraction) or Conventional Fractionated Radiotherapy: 50-70 Gy total (1.8-2.5 Gy/fraction).Dose determined by investigator. Immunotherapy Phase: Iparomlimab and Tuvonralimab: Dose: 5 mg/kg IV every 3 weeks (Day 1). Infusion: Diluted in 100 mL saline/5% glucose, administered over 20-60 minutes. Duration: Until disease progression, intolerable toxicity, new antitumor therapy, or up to 1 year. Progression Management: Continuation post-progression permitted after investigator-patient discussion; permanent discontinuation upon re-progression.
  Interventions: Combination Product: Spatially Fractionated Radiation Therapy Followed by Sequential Hypofractionated or Conventional Fractionated Radiotherapy Combined with Iparomlimab and Tuvonralimab

INTERVENTIONS:
Combination Product: Spatially Fractionated Radiation Therapy Followed by Sequential Hypofractionated or Conventional Fractionated Radiotherapy Combined with Iparomlimab and Tuvonralimab — Radiotherapy Phase: Spatially fractionated radiotherapy (SFRT, 10-20 Gy/1F) to the tumor, followed by hypofractionated/conventional fractionated radiotherapy (dose investigator-determined).
  Immunotherapy Phase: Iparomlimab and Tuvonralimab (5 mg/kg) initiated within 1 week post-radiotherapy, infused IV over 20-60 minutes (Day 1, every 3 weeks) in 100 mL saline/5% glucose. Treatment continues until disease progression, intolerable toxicity, new antitumor therapy, consent withdrawal, or investigator decision, with a maximum duration of 1 year. Progression may allow continued therapy after patient-investigator discussion; re-progression mandates permanent discontinuation.

SUMMARY:
Study Objectives Primary Objective:To evaluate the safety of SFRT followed by hypofractionated/conventional fractionated radiotherapy combined with Iparomlimab and Tuvonralimab Injection in relapsed/refractory bulky solid tumors.

Secondary Objectives:To assess efficacy (objective response rate, disease control rate, progression-free survival, etc.) and identify predictive biomarkers.To explore correlations between immunologic biomarkers (e.g., PD-L1 expression, plasma IL-2/IL-10) and treatment outcomes.

Study Endpoints Primary: Safety (incidence/severity of treatment-related adverse events).

Secondary:

ORR, DCR, DoR, mPFS, mOS Exploratory: Biomarker analysis (PD-L1, IL-2, IL-10).

DETAILED DESCRIPTION:
1. Study Title A Study of Spatially Fractionated Radiation Therapy Followed by Sequential Hypofractionated or Conventional Fractionated RT Combined with Iparomlimab and Tuvonralimab for Relapsed and Refractory Bulky Solid Tumors
2. Study Objectives Primary Objective: To evaluate the safety of SFRT followed by hypofractionated/Conventional Fractionated radiotherapy combined with Iparomlimab and Tuvonralimab in relapsed/refractory bulky solid tumors.

   Secondary Objectives:

   To assess efficacy (objective response rate, disease control rate, progression-free survival, etc.) and identify predictive biomarkers.To explore correlations between immunologic biomarkers (e.g., PD-L1 expression, plasma IL-2/IL-10) and treatment outcomes.
3. Study Design Type: Prospective, single-arm, open-label, single-center clinical study. Target Population: Patients with relapsed/refractory bulky solid tumors (≥6 cm in diameter).

   Sample Size: 30 participants (based on primary safety endpoint).
4. Patient Selection

   Inclusion Criteria:

   Age 18-75 years. Histologically confirmed malignancy with post-treatment recurrence (local or metastatic).

   At least one measurable lesion (>6 cm) unsuitable for surgery/ablation. ECOG performance status 0-2; life expectancy ≥3 months.

   Adequate organ function (within 14 days prior to enrollment):

   ANC ≥1.5×10⁹/L; platelets ≥90×10⁹/L; hemoglobin ≥8 g/dL. Serum albumin ≥2.8 g/dL; total bilirubin ≤1.5×ULN; ALT/AST ≤2.5×ULN (≤5×ULN with liver metastases).

   Creatinine ≤1.5×ULN or CrCl ≥60 mL/min. INR/APTT ≤1.5×ULN (stable anticoagulation allowed). Negative pregnancy test (for women of childbearing potential). Willingness to comply with protocol and provide informed consent.

   Exclusion Criteria:

   Severe hypersensitivity to study drugs. History of cardiovascular events (e.g., myocardial infarction, stroke) within 6 months.

   Active autoimmune disease (exceptions: controlled type 1 diabetes, hypothyroidism, localized skin conditions).

   Immunodeficiency (e.g., HIV, organ transplant). Systemic corticosteroids (>10 mg prednisone equivalent/day) within 2 weeks prior to treatment.

   Pregnancy, lactation, or refusal to use contraception. Other conditions deemed unsuitable by the investigator.
5. Treatment Protocol

Radiotherapy Phase:

SFRT: 10-20 Gy/1 fraction to the tumor. Sequential Radiotherapy:Hypofractionated Radiotherapy: 20-70 Gy total (3-12.5 Gy/fraction) or Conventional Radiotherapy: 50-70 Gy total (1.8-2.5 Gy/fraction).Dose determined by investigator.

Immunotherapy Phase:

Iparomlimab and Tuvonralimab:

Dose: 5 mg/kg IV every 3 weeks (Day 1). Infusion: Diluted in 100 mL saline/5% glucose, administered over 20-60 minutes. Duration: Until disease progression, intolerable toxicity, new antitumor therapy, or up to 1 year.

Progression Management: Continuation post-progression permitted after investigator-patient discussion; permanent discontinuation upon re-progression.

6. Study Endpoints

1. Primary Endpoint(s) & Definitions Safety Evaluation: Adverse events (treatment-related toxicities) assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.
2. Secondary Endpoints & Definitions

   1. Complete Response (CR) Rate: Defined as the proportion of patients achieving complete response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
   2. Objective Response Rate (ORR): The proportion of patients achieving a reduction in tumor size meeting predefined criteria (Complete Response [CR]: disappearance of all target lesions; Partial Response [PR]: ≥30% reduction in the sum of target lesion diameters) per RECIST V1.1, sustained for a minimum duration.
   3. Disease Control Rate (DCR): Defined as the proportion of patients achieving tumor response (partial response [PR] + complete response [CR]) or stable disease (SD) per RECIST v1.1, sustained for a minimum required duration.
   4. Duration of Response (DoR): The time from achieving an objective response (CR or PR) to disease progression or recurrence. For example, in lung cancer targeted therapy trials, DoR measures the interval from achieving PR to tumor regrowth or new lesion development.
   5. Median Progression-Free Survival (mPFS): Defined as the median time from treatment initiation to the first documented disease progression or death from any cause, whichever occurs first.
   6. Median Overall Survival (mOS): Defined as the median time from treatment initiation to death from any cause.

      7.Statistical Analysis Descriptive statistics for demographics, efficacy, and safety data. Kaplan-Meier method for survival analysis (mOS, mPFS). 95% confidence intervals for response rates. AE reporting: Incidence, severity, causality, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female.
2. Histologically confirmed malignant tumor in the past.
3. Disease recurrence after treatment, including local regional relapsed and distant metastasis.
4. At least one measurable lesion with a maximum diameter greater than 6 cm, unsuitable for conventional surgery, ablation, or other treatments.
5. ECOG: 0-2 points.
6. Expected survival ≥3 months.
7. Washout period of previous anti-tumor treatment >4 weeks.
8. The patient agrees and signs the informed consent form.
9. The function of vital organs meets the following requirements (no use of any blood components, cell growth factors, leukocyte boosters, platelet boosters, or anemia correction drugs within 14 days prior to the first use of the study drug):

   1. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
   2. Platelets ≥90×10^9/L;
   3. Hemoglobin ≥8g/dL;
   4. Serum albumin ≥2.8g/dL;
   5. Total bilirubin ≤1.5×ULN, ALT, AST, and/or AKP ≤2.5×ULN; if liver metastasis is present, ALT and/or AST ≤5×ULN; if liver or bone metastasis is present, AKP ≤5×ULN;
   6. Serum creatinine ≤1.5×ULN or creatinine clearance rate greater than 60 mL/min;
   7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5×ULN (patients on stable doses of anticoagulation therapy such as low molecular weight heparin or warfarin with INR within the expected therapeutic range can be screened).
10. Negative pregnancy test for female subjects (for female patients of childbearing potential);
11. The subject voluntarily joins the study, signs the informed consent form, has good compliance, and cooperates with follow-up;
12. The investigator believes that the patient may benefit.

Exclusion Criteria:

1. History of severe immediate hypersensitivity reaction to any of the drugs used in this study.
2. Any of the following conditions within 6 months prior to screening: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism. Patients known to have coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be on an optimized stable medical regimen as determined by the treating physician; consultation with a cardiologist may be appropriate if necessary.
3. History of receiving anti-tumor vaccines or live vaccines within 4 weeks prior to the first dose of the investigational drug.
4. Active autoimmune diseases or history of autoimmune diseases that may recur. However, patients with the following conditions are not excluded and can proceed to further screening:

   1. Controlled Type 1 diabetes
   2. Hypothyroidism (if it can be controlled with hormone replacement therapy alone)
   3. Skin conditions that do not require systemic therapy (e.g., vitiligo, psoriasis, alopecia)
   4. Any other condition not expected to recur without external triggering factors
5. Lack of civil capacity or limited civil capacity.
6. Physical or mental conditions that impair the patient's ability to fully or adequately understand the potential complications of this study, as judged by the investigator.
7. Patients with an expected survival of less than 3 months.
8. Patients with significantly diminished cardiac, hepatic, pulmonary, renal, and bone marrow function.
9. Drug abuse or alcohol addiction.
10. Tumor lesions invading major blood vessels such as the internal carotid artery and vein and their major branches, posing a high risk of bleeding.
11. Subjects requiring systemic treatment with corticosteroids (more than 10mg/day prednisone equivalent dose) or other immunosuppressive agents within 2 weeks prior to the first use of the investigational drug, except for the use of corticosteroids for local esophageal inflammation and prevention of allergies and nausea/vomiting. Special cases need to be discussed with the sponsor. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal corticosteroid replacements at doses >10mg/day prednisone equivalent are allowed.
12. History of immunodeficiency, including HIV-positive status, or other acquired or congenital immunodeficiency disorders, or history of organ transplantation or allogeneic bone marrow transplantation.
13. Pregnant or breastfeeding female patients, male or female patients of childbearing potential who are unwilling or unable to use contraception for at least 1 year after the end of the treatment protocol throughout the study period.
14. The investigator deems the patient unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2028-06-19 (Estimated); Study Completion 2029-06-19 (Estimated)

PRIMARY OUTCOMES:
Safety (treatment-related toxicity and adverse reactions) | The safety endpoints will be assessed by a review of adverse events and serious adverse events according to CTCAE up to 1 year after end of treatment
  Adverse events (treatment toxicity) will be evaluated using NCI-CTCAE version 5.0.

SECONDARY OUTCOMES:
Complete Response (CR) rate | One imageological examination will be performed during the baseline period, followed by another imageological examination after the completion of radiotherapy. During immunotherapy, imaging assessments will be conducted every 3 treatment cycles.
  Complete Response (CR) rate assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of Response (DoR) | One imageological examination will be performed during the baseline period, followed by another imageological examination after the completion of radiotherapy. During immunotherapy, imaging assessments will be conducted every 3 treatment cycles.
  Duration of Response (DoR) refers to the time from when a patient first achieves a complete response or partial response until disease progression or death due to any cause.
Objective Response Rate (ORR) | One imageological examination will be performed during the baseline period, followed by another imageological examination after the completion of radiotherapy. During immunotherapy, imaging assessments will be conducted every 3 treatment cycles.
  Objective Response Rate (ORR) refers to the proportion of patients who achieve a best overall response of complete or partial response according to the RECIST 1.1 criteria.
Median Progression-Free Survival (mPFS) | One imageological examination will be performed during the baseline period, followed by another imageological examination after the completion of radiotherapy. During immunotherapy, imaging assessments will be conducted every 3 treatment cycles.
  Median Progression-Free Survival (mPFS) refers to the median time from the start of treatment until the first discovery of disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | One imageological examination will be performed during the baseline period, followed by another imageological examination after the completion of radiotherapy. During immunotherapy, imaging assessments will be conducted every 3 treatment cycles.
  Disease Control Rate (DCR) refers to the proportion of patients who achieve a response of partial response (PR) or complete response (CR) and those who have stable disease (SD) lasting for at least a minimum duration requirement, as per the RECIST 1.1 criteria for solid tumors.
Median Overall Survival (mOS) | One imageological examination will be performed during the baseline period, followed by another imageological examination after the completion of radiotherapy. During immunotherapy, imaging assessments will be conducted every 3 treatment cycles.
  Median Overall Survival (mOS) refers to the median time from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Anwen Liu, Ph.D., Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No